CLINICAL TRIAL: NCT01771042
Title: Neuroadrenergic Dysfunction Along the Diabetes Continuum: Benefits of Weight Loss Within Different Strata of Metabolic Risk
Brief Title: The Effects of Weight Loss on Neuroadrenergic Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Baker Heart Research Institute (Other)
Responsible Party: Principal Investigator, Nora E. Straznicky, Group Leader/Senior Research Officer, Baker Heart Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/13; 1/13 (Other Grant/Funding Number: Diabetes Australia Millenium Grant)
Record Dates: First submitted 2013-01-15; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Obesity; Type 2 Diabetes; Metabolic Syndrome
Keywords: weight loss; metabolic syndrome; sympathetic nervous system; insulin resistance; glucose tolerance
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Metabolic Syndrome; Weight Loss; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal glucose tolerant (Experimental): Weight loss attained by 25% caloric restriction.
  This arm will be both a glycemic and time control. Initially they will undergo a 4-month weight maintenance phase (acting as time control), followed by 4 month weight loss.
  Interventions: Other: Dietary weight loss at 25% energy deficit
- Impaired glucose tolerant (Experimental): Weight loss using 25% caloric restriction.
  Impaired glucose tolerant subjects will undergo 4 months weight loss (25% caloric deficit) followed by 3 months weight loss maintenance
  Interventions: Other: Dietary weight loss at 25% energy deficit
- Type 2 diabetic hyperinsulinemic (Experimental): Weight loss using 25% caloric restriction.
  This group will undergo 4 months weight loss (25% caloric deficit) followed by 3 months weight loss maintenance
  Interventions: Other: Dietary weight loss at 25% energy deficit
- Type 2 diabetic hypoinsulinemic (Experimental): Weight loss via 25% caloric restriction.
  This group will undergo 4 months weight loss (25% caloric deficit) followed by 3 months weight loss maintenance
  Interventions: Other: Dietary weight loss at 25% energy deficit

INTERVENTIONS:
Other: Dietary weight loss at 25% energy deficit — Dietary weight loss at 25% energy deficit. Dietary macronutrient content will comprise 25% protein, 30% fat and 45% carbohydrate.

SUMMARY:
Elevated subconscious nervous system activity is a characteristic of the obese state and contributes importantly to the risk of heart disease and diabetes. This project will compare sympathetic nervous system activity and function in a group of obese persons with differing levels of sugar tolerance (normal, impaired and type 2 diabetic). Inter-relationships with insulin action, blood pressure, heart and kidney function will be determined before and after a 4-month weight loss and 3-month weight loss maintenance program.

It is hypothesized that the transition from normal sugar tolerance to impaired sugar tolerance to type 2 diabetes will be accompanied by escalating sympathetic nervous system dysfunction. Furthermore, that weight loss will favorably improve sympathetic function, with greatest benefits occurring in those subjects who are insulin resistant with high blood insulin concentration.

DETAILED DESCRIPTION:
The twin epidemics of obesity and diabetes represent a major public health problem worldwide. There is a growing body of evidence to suggest that autonomic dysfunction, comprising elevated sympathetic nervous system (SNS) activity and blunted sympathetic neural responsiveness plays a role in both the pathogenesis and target organ complications of obesity and diabetes. The proposed project will undertake a detailed comparative analysis of neuroadrenergic function along the diabetes continuum, its inter-relationship with insulin sensitivity and secretion, and target organ function, and the benefits of active weight loss and weight loss maintenance within different strata of metabolic risk.

ELIGIBILITY:
Inclusion Criteria:

Men and postmenopausal women (n=120), untreated, weight-stable, non-smoking, aged 45-65 years, BMI 27-45 kg/m2, will be recruited. Glucose tolerance status will be determined by a 75-g oral glucose tolerance test (OGTT), using WHO criteria (53): normal glucose tolerance, fasting plasma glucose < 7.0 mmol/L and 2-h plasma glucose < 7.8 mmol/L; IGT, fasting plasma glucose < 7.0 mmol/L and 2-h plasma glucose > 7.8 and < 11.1 mmol/L; T2D, fasting plasma glucose > 7.0 mmol/L or 2-h plasma glucose > 11.1 mmol/L. Hyper-insulinemia will be defined as an insulin area under the curve during OGTT > 8000 mU/L ∙ min-1 and hypo-insulinemia as < 8000 mU/L ∙ min-1.

Exclusion Criteria:

Prior history of cardiovascular disease (previous myocardial infarction, angina, stroke, heart failure, secondary hypertension), renal (serum creatinine >0.12 mmol/L or estimated GFR <60 ml/min/1.73 m2) or hepatic disease or diseases which may affect measured parameters (e.g. thyroid disease); severe hypertension; a history of surgical weight loss; CPAP therapy; and >4 alcoholic drinks/day. T2D individuals with moderate hyperglycemia (HbA1c >9%) will be excluded so that hypoglycaemic pharmacotherapy may be instituted (54). Participants will be sought through newspaper advertising and poster displays in primary health care centres (General Practices). Newly diagnosed T2D subjects

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Change in whole-body norepinephrine kinetics | 4 months and 7 months
  The study will examine the dynamic processes of norepinephrine spillover into and removal from the central plasma compartment using the isotope dilution technique.Measurements will be made at baseline, after 4 months active weight loss, and again after 3 months weight loss maintenance. The weight loss maintenance phase will permit differentiation of the effects of active weight loss (incorporating both negative energy balance and weight loss per se) and stable lower body weight on sympathetic neural parameters.

SECONDARY OUTCOMES:
Change in muscle sympathetic nerve activity | 4 months and 7 months
  Muscle sympathetic nerve firing will be quantified by the technique of mirconeurography at baseline and after 4 months active weight loss and 3 months weight loss maintenance. The weight loss maintenance phase will permit differentiation of the effects of active weight loss (incorporating both negative energy balance and weight loss per se) and stable lower body weight on sympathetic nerve firing and pattern.

OTHER OUTCOMES:
Change in insulin sensitivity | 4 months and 7 months
  Insulin sensitivity will be assessed by the gold standard euglycemic hyperinsulinemic clamp method at baseline and after 4 months active weight loss and 3 months weight loss maintenance. The weight loss maintenance phase will permit differentiation of the effects of active weight loss (incorporating both negative energy balance and weight loss per se) and stable lower body weight on insulin sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nora E Straznicky, PhD MPH, Principal Investigator — Baker IDI Heart & Diabetes Institute
Locations (1):
- Baker IDI Heart & Diabetes Institute, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Straznicky NE, Grima MT, Sari CI, Lambert EA, Phillips SE, Eikelis N, Kobayashi D, Hering D, Mariani JA, Dixon JB, Nestel PJ, Karapanagiotidis S, Schlaich MP, Lambert GW. Reduction in peripheral vascular resistance predicts improvement in insulin clearance following weight loss. Cardiovasc Diabetol. 2015 Aug 22;14:113. doi: 10.1186/s12933-015-0276-2. PMID 26297500
- [Derived] Straznicky NE, Grima MT, Lambert EA, Sari CI, Eikelis N, Nestel PJ, Phillips SE, Hering D, Karapanagiotidis S, Dixon JB, Schlaich MP, Lambert GW. Arterial norepinephrine concentration is inversely and independently associated with insulin clearance in obese individuals with metabolic syndrome. J Clin Endocrinol Metab. 2015 Apr;100(4):1544-50. doi: 10.1210/jc.2014-3796. Epub 2015 Jan 15. PMID 25590214